CLINICAL TRIAL: NCT00242281
Title: A Phase III, Multicenter Study to Evaluate the Safety/Efficacy of APC-111 MP Tablet QD vs. Penicillin VK QID Both for 10 Days Treatment of Pharyngitis Secondary to S.Pyogenes in Adolescents/Adults
Brief Title: APC-111 MP Tablet Once a Day vs.Penicillin VK Four Times a Day Both for 10 Days in Patients With Strep Throat
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Advancis Pharmaceutical Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111.302
Record Dates: First submitted 2005-10-18; First posted 2005-10-20 (Estimated); Last update posted 2006-10-25 (Estimated); Status verified 2006-01

CONDITIONS: Sore Throat; Pharyngitis; Tonsillitis
Keywords: Sore Throat; Pharyngitis; Tonsillitis
MeSH Terms: conditions — Pharyngitis; Tonsillitis

INTERVENTIONS:
Drug: APC-111 MP Tablet, 775 mg

SUMMARY:
The primary objective of this study is to evaluate the efficacy of APC 111 MP Tablet, 775 mg tablet, given orally (PO)once daily (QD) for 10 days compared to that of Penicillin VK, 250 mg PO four times daily (QID) for 10 days in terms of bacteriological outcome at the Test-of-Cure (TOC) Visit (Day 14-18) in the eligible Per-Protocol bacteriological (PPb) population.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent/assent
* Age 12 and older
* A clinical diagnosis of acute tonsillitis and/or pharyngitis defined as having the clinical signs and symptoms compatible with tonsillitis and/or pharyngitis, including sore throat and pharyngeal erythema with at least one of the following:

  * Odynophagia
  * Tonsillar or pharyngeal exudates
  * Tender cervical lymph nodes
  * Fever or history of fever treated with antipyretics
  * Chills
  * Uvular edema
  * Elevated white blood cell count
  * Red tongue and prominent papillae
* A positive rapid screening test for S. pyogenes
* Subject is an appropriate candidate for oral antibiotic therapy and can swallow the study dosage forms
* Females must be non-lactating and:

  * At no risk of pregnancy for one of the following reasons: post-menopausal for at least one year, hysterectomy, tubal ligation, or abstinent from sexual activity that could result in pregnancy, OR
  * If of child-bearing potential and sexually active, the patient must have a negative baseline urine pregnancy test and be utilizing acceptable contraceptives throughout the study.
  * If of child bearing potential and not currently sexually active, the patient must have a negative baseline urine pregnancy test and must agree to remain abstinent for the duration of the study. If they decide to become sexually active during the period of the study, they must agree to use acceptable contraception.
* Are able to comply with the requirements of the protocol

Exclusion Criteria:

* Chronic or recurrent odynophagia or enlarged tonsils of obscure etiology
* More than one episode of acute tonsillitis and/or pharyngitis in the 6 months prior to baseline visit
* Pharyngitis known or suspected to be due to a pathogen resistant to β-lactam antimicrobials
* Subjects who are known carriers of S. pyogenes
* Previous allergies, serious adverse reaction to, or intolerance to penicillin or any other member of the β-lactam class of antimicrobials, including cephalosporins
* Any serious illness or concomitant condition that the Investigator judges would preclude the study evaluations or make it unlikely that the course of study therapy and follow-up could be completed. This would also include:

  * Any rapidly progressive underlying disease with a shortened life expectancy
  * The inability to swallow the study dosage form
  * Unable to understand the requirements of the study
  * Neutropenia (<1000 PMNs/mm3) or other immunocompromised state.
* Concurrent condition of upper/lower respiratory tract infections
* Concurrent symptoms of viral etiology including:

  * conjunctivitis, coryza, and cough
  * diffuse adenopathy or rash suggestive of mononucleosis
  * rash or arthropathy suggestive of scarlet fever
* Seizure disorder, lowered seizure threshold, or psychiatric condition requiring use of major tranquilizers
* Pregnancy or nursing
* Expectation that additional effective systemic antibacterials would be required for any condition during the duration of the study
* Current drug or alcohol abuse
* Receipt of any experimental drug or medical device within the previous 30 days
* Previous treatment under this protocol
* The need for hospitalization or I.V. antimicrobial therapy
* Previous systemic antimicrobial therapy within 30 days
* The presence of clinically significant hematologic conditions
* History of cardiovascular disease, renal disease, or neurological disease secondary to previous infection with S. pyogenes or previous rheumatic fever
* Probenecid treatment or systemic steroids for 7 days prior to baseline visit and throughout the duration of the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600
Dates: Start 2005-11; Study Completion 2006-07

PRIMARY OUTCOMES:
The bacteriological outcome at the Test - of - Cure Visit (Day 14-18)

SECONDARY OUTCOMES:
The bacteriological outcome at the Late Post Therapy visit (Day 38-45)
Clinical Outcome at TOC and LPT
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Susan P Clausen, PhD, Study Director — Advancis Pharmaceutical Corp
Locations (41):
- United States (35):
  - Birmingham, Alabama
  - Tallassee, Alabama
  - Phoenix, Arizona
  - Carmichael, California
  - Laguna Niguel, California
  - San Luis Obispo, California
  - Littleton, Colorado
  - DeLand, Florida
  - Conyers, Georgia
  - Boise, Idaho
  - Overland Park, Kansas
  - Topeka, Kansas
  - Wichitia, Kansas
  - Bardstown, Kentucky
  - Milford, Massachusetts
  - New Bedford, Massachusetts
  - Kalamazoo, Michigan
  - Butte, Montana
  - Omaha, Nebraska
  - Johnson City, New York
  - Burlington, North Carolina
  - Simpsonville, North Carolina
  - Canfield, Ohio
  - North Wales, Pennsylvania
  - Scotland, Pennsylvania
  - Shippensburg, Pennsylvania
  - Bristol, Tennessee
  - Kingsport, Tennessee
  - San Antonio, Texas
  - Bountiful, Utah
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Newport News, Virginia
  - Edmonds, Washington
  - Wenatchee, Washington
- Canada (6):
  - Coquitlam, British Columbia
  - Fort Erie, Ontario
  - Markham, Ontario
  - Toronto, Ontario
  - Saint-Jermone, Quebec
  - Sherbrooke, Quebec